CLINICAL TRIAL: NCT00975390
Title: The Effect of Caffeine or Protein Co-ingestion With Carbohydrate on Post-exercise Muscle Glycogen Synthesis Rate.
Brief Title: Muscle Glycogen Synthesis When Caffeine and Protein is Co-Ingested With Carbohydrates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Milou Beelen, Dr., Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 08-3-066
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Exercise Recovery
Keywords: Glycogen; Carbohydrate; Protein; Caffeine; Post exercise muscle glycogen synthesis; Sports nutrition
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Carbohydrate ingestion
  Interventions: Dietary Supplement: Carbohydrate
- 2 (Experimental): Carbohydrate and protein ingestion
  Interventions: Dietary Supplement: Carbohydrate and protein ingestion
- 3 (Experimental): Carbohydrate and caffeine ingestion
  Interventions: Dietary Supplement: Carbohydrate and caffeine ingestion

INTERVENTIONS:
Dietary Supplement: Carbohydrate — 1.2 g/kg/h
  Arms: 1
Dietary Supplement: Carbohydrate and protein ingestion — 1.2 g/kg/h carbohydrate plus 0.4 g/kg/h protein
  Arms: 2
Dietary Supplement: Carbohydrate and caffeine ingestion — 1.2 g/kg/h carbohydrate and 1.67 g/kg/h caffeine
  Arms: 3

SUMMARY:
The aim of the present study is to investigate the effect of added protein+leucine or caffeine to 1.2 g/kg/h CHO on the rate of post-exercise muscle glycogen re-synthesis in healthy, recreational athletes.

The investigators hypothesize that both interventions (the addition of caffeine or protein+leucine) will lead to higher glycogen re-synthesis compared to the ingestion of CHO only, and that the co-ingestion of protein and leucine will result in the highest muscle glycogen synthesis rates.

ELIGIBILITY:
Inclusion Criteria:

* male cyclists
* healthy
* BMI < 25

Exclusion Criteria:

* female
* use of medication
* non cycling
* BMI > 25

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Muscle glycogen synthesis rates | 6 hours

SECONDARY OUTCOMES:
Glycogen synthase activity, plasma glucose, insulin, free fatty acids and epinephrine responses | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands